CLINICAL TRIAL: NCT04455308
Title: Chilblains, COVID-19 and Lockdown: Epidemiologic Study
Brief Title: COVID-19 and Chilblains
Acronym: ECCES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC20_8888_ECCES
Record Dates: First submitted 2020-06-30; First posted 2020-07-02 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2023-05

CONDITIONS: Chilblains; COVID-19
MeSH Terms: conditions — Chilblains; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects with chilblains (Experimental)
  Interventions: Other: Biological sample collection
- Subjects without chilblains (Active Comparator)
  Interventions: Other: Biological sample collection

INTERVENTIONS:
Other: Biological sample collection — 10mL blood sample

SUMMARY:
Chilblains (inflammatory lesion of the feet or hands) have been reported with an unusual frequency during the confinement period, most commonly in children, teenagers and young adults. The aim of the ECCES study is to find out whether these manifestations of chilblains can be linked to the SARS-CoV-2 coronavirus.

For this, an epidemiologic study will compare two types of family (or more precisely people who were confined together in March-April-May):

* "case family" in which at least one of the members had chilblains
* "comparator family" in which none of the members had chilblains Environment (home lockdown) of the two types of family will be analyzed. Each member of the "family" will be suggested doing a serological test.

ELIGIBILITY:
Inclusion Criteria:

* "case family"
* at least one of the members with chilblains
* diagnosis of chilblains (anamnesis and pictures) written informed consent
* "comparator family"
* none of the members with chilblains
* one member matched on age (+/- 1 year) to a patient with chilblains
* written informed consent

Exclusion Criteria:

- Subject legally protected (under judicial protection, guardianship), persons deprived of liberty

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-10-19 (Actual)

PRIMARY OUTCOMES:
Level of viral exposure in "case family" compared to "comparator family" | Through study completion, an average of 3 months

SECONDARY OUTCOMES:
Comparison of seropositivity rates in subjects with chilblains and their age-matched controls | Through study completion, an average of 3 months
Comparison of SARS-CoV-2 seropositivity rates among members of case (subject with chilblains) and control (subject without chilblains) outbreaks | Through study completion, an average of 3 months
Antibody avidity and differentiated IgG and IgM assay by subject in the homes | Through study completion, an average of 3 months

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU Angers, Angers
  - CHRU Brest, Brest
  - CHU Nantes, Nantes
  - CHU Rennes, Rennes
  - CHRU Tours, Tours

REFERENCES:
- [Result] Poizeau F, Barbarot S, Le Corre Y, Brenaut E, Samimi M, Aubert H, Toubel A, Dupuy A. Long-term Outcome of Chilblains Associated with SARS-CoV-2. Acta Derm Venereol. 2021 Dec 13;101(12):adv00614. doi: 10.2340/00015555-3930. PMID 34515805
- [Result] Poizeau F, Oger E, Barbarot S, Le Corre Y, Samimi M, Brenaut E, Aubert H, Chambrelan E, Droitcourt C, Gissot V, Heslan C, Laurent C, Martin L, Misery L, Tattevin P, Toubel A, Thibault V, Dupuy A. Chilblains during lockdown are associated with household exposure to SARS-CoV-2: a multicentre case-control study. Clin Microbiol Infect. 2022 Feb;28(2):285-291. doi: 10.1016/j.cmi.2021.09.032. Epub 2021 Oct 4. PMID 34619397